CLINICAL TRIAL: NCT06535165
Title: Effect of 14-day Red Beetroot Juice Intake on Physical Function, Gut Microbiota Composition, and Systemic Inflammation in Adults With Long COVID-19
Brief Title: Effect of Red Beetroot Juice Intake in Adults With Long COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesco Landi, MD, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 5110
Record Dates: First submitted 2024-08-01; First posted 2024-08-02 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red Beetroot Juice (Experimental): daily oral supplementation with 200 mL beetroot juice for 14 days
  Interventions: Dietary Supplement: Red Beetroot Juice
- Control (Placebo Comparator): Placebo (a solution containing 7 g of sugar, 180 mL of water, and 20 mL of beetroot juice, to show the same color as the active treatment) for 14 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Red Beetroot Juice — 200ml/d for 14 days
  Arms: Red Beetroot Juice
Other: Placebo — 200ml/d for 14 days
  Arms: Control

SUMMARY:
Red beetroot juice may have positive effects on multiple pathways involved in long COVID. The aim of this pilot study was to explore the impact of beetroot juice supplementation on physical function, gut microbiota, and systemic inflammation in adults with long-COVID

DETAILED DESCRIPTION:
A single-center, double-blind, placebo-controlled randomized trial to test the effects of 14 days of beetroot juice supplementation on functional and biological outcomes in adults with long-COVID.

Participants were randomized 1:1 to receive either daily oral supplementation with 200 mL beetroot juice or placebo for 14 days. The primary endpoint was the change from baseline to day 14 in the fatigue resistance test. Secondary outcomes included the distance walked on the 6-min walk test, handgrip strength, and flow-mediated dilation. Secondary endpoints also included changes from baseline in circulating inflammatory mediators, metagenomic and fecal water metabolomic profiles. Partial least squares discriminant analysis (PLS-DA) models were built to evaluate the differences in biological variables associated with the interventions.

ELIGIBILITY:
Inclusion Criteria:

* a certification of a previous SARS-CoV-2 infection
* a negative COVID-19 swab test at least four weeks prior to the screening visit
* meet the criteria for long-COVID diagnosis according to the World Health Organization criteria
* report persistent fatigue

Exclusion Criteria:

* intolerance to beetroot juice or its derivatives
* clinical conditions and/or use of medications that may interfere with trial outcomes (e.g., pregnancy or breastfeeding, diabetes, use of steroids or non-steroidal anti-inflammatory drugs, immunosuppressants, nitrates)
* participation in other intervention trials for long-COVID

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Fatigue resistance | 14 days
  The time (in seconds) when the pressure dropped to 50% of the maximum grip strength

SECONDARY OUTCOMES:
Six-minute walk test | 14 days
  The distance walked (in meters) on the 6-min walk test
Flow-mediated dilation | 14 days
  the dilation of the brachial artery after a transitory bout of forearm ischemia
Changes in the concentration of gut microbial species | 14 days
  Changes in the concentration of gut microbial species as assessed through 16S rRNA analysis
Fecal water metabolomics | 14 days
  Changes in fecal water metabolomics by nuclear magnetic resonance (NMR) spectroscopy
Changes in the concentration of circulating inflammatory mediators | 14 days
  Changes in the concentration of circulating cytokines, chemokines, growth factors, extracellular vesicles

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Landi, MD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Center for Aging and Geriatrics Research - UCSC, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Calvani R, Giampaoli O, Marini F, Del Chierico F, De Rosa M, Conta G, Sciubba F, Tosato M, Picca A, Ciciarello F, Galluzzo V, Gervasoni J, Di Mario C, Santoro L, Tolusso B, Spagnoli M, Tomassini A, Aureli W, Toto F, Pane S, Putignani L, Miccheli A, Marzetti E, Landi F; Gemelli against COVID-19 Post-Acute Care Team. Beetroot juice intake positively influenced gut microbiota and inflammation but failed to improve functional outcomes in adults with long COVID: A pilot randomized controlled trial. Clin Nutr. 2024 Dec;43(12):344-358. doi: 10.1016/j.clnu.2024.11.023. Epub 2024 Nov 14. PMID 39571342